CLINICAL TRIAL: NCT05972720
Title: An Open-label, Multicenter Phase 2 Study Evaluating the Efficacy and Safety of Firi-cel, a CD22-directed Autologous Chimeric Antigen Receptor (CAR) T-cell Therapy in Patients With Relapsed/Refractory Large B-Cell Lymphoma After CD19-directed CAR T-cell Therapy
Brief Title: A Phase 2 Study of Firi-cel in Patients With Relapsed/Refractory Large B-cell Lymphoma
Acronym: FIRCE-1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision to stop trial, withdraw the IND and close down operations.
Sponsor: CARGO Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRG-022-101
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Cancer; Relapsed/Refractory Large B-cell Lymphoma (LBCL)
Keywords: Lymphoma; CD-22 Expressing Tumor; Chimeric Antigen Receptor; Adoptive Immunotherapy; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Primary Mediastinal B-cell; Lymphoma, Transformed; Lymphoma, Transformed Non-Hodgkin; Lymphoma, Non-Hodgkin; CAR T; CAR T-cell therapy; Cell Therapy; Cellular Immuno-therapy; CRG-022; CD22; FIRCE-1; firicabtagene autoleucel; firi-cel
MeSH Terms: conditions — Neoplasms; Recurrence; Lymphoma; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin | interventions — fludarabine; Cyclophosphamide; Drugs, Investigational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental Drug (Cohort 1) (Experimental): Single infusion of firi-cel following conditioning chemotherapy
  Interventions: Drug: Fludarabine (Conditional therapy); Drug: Cyclophosphamide Monohydrate (Conditional therapy); Drug: firi-cel (Experimental drug)
- Experimental Drug (Cohort 2: non-conforming product) (Experimental): Single infusion of firi-cel following conditioning chemotherapy (patients in this cohort will receive non-conforming firi-cel that is deemed safe to administer).
  Interventions: Drug: Fludarabine (Conditional therapy); Drug: Cyclophosphamide Monohydrate (Conditional therapy); Drug: firi-cel (Experimental drug)
- Experimental Drug (Cohort 3) (Experimental): Patients with relapsed or refractory Large B-cell lymphoma who have previously been treated with bispecific T-cell engaging antibody therapy will receive a single infusion of firi-cel following conditioning chemotherapy.
  Interventions: Drug: Fludarabine (Conditional therapy); Drug: Cyclophosphamide Monohydrate (Conditional therapy); Drug: firi-cel (Experimental drug)

INTERVENTIONS:
Drug: Fludarabine (Conditional therapy) — Lymphodepletion chemotherapy
Drug: Cyclophosphamide Monohydrate (Conditional therapy) — Lymphodepletion chemotherapy
Drug: firi-cel (Experimental drug) — Investigational agent

SUMMARY:
This is a prospective, open-label, multi-center clinical study designed to evaluate the safety, tolerability, efficacy, pharmacokinetics, pharmacodynamics, and immunogenicity of firicabtagene autoleucel (firi-cel), a CD22-directed autologous Chimeric Antigen Receptor (CAR) T-cell therapy for the treatment of relapsed or refractory large B-cell lymphoma (LBCL).

DETAILED DESCRIPTION:
Firicabtagene autoleucel (firi-cel) is an autologous CAR T-cell therapy targeting CD22, a common B-cell antigen widely expressed in LBCL. This Phase 2 study is designed to evaluate the safety and the efficacy of firi-cel in patients with R/R LBCL that has progressed after CD19-directed CAR T-cell therapy. The study is designed to treat up to 123 patients with a single infusion of firi-cel.

ELIGIBILITY:
Key Inclusion Criteria:

* Aged ≥18 years
* Relapsed or refractory, histologically confirmed large B-cell lymphoma.
* Must have relapsed or refractory diseae after last therapy.
* For enrollment in cohort 1, patients must have previously received a CD19-directed CAR T-cell therapy
* For enrollment in cohort 3, patients must have received at least two prior lines of therapy including a bispecific T-cel engaging antibody therapy.
* Must have at least one radiographically measurable lesion.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate hematological, renal, and liver function
* Willing and able to remain within 1 hour of the treating center for at least 4 weeks after infusion.

Key Exclusion Criteria:

* Clinically significant concurrent medical illness
* Active fungal, bacterial, viral or other infection.
* Prior allogeneic stem cell transplant or allogeneic cell therapy

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Objective response rate - Blinded independent review | Up to 24 months
  Percentage of patients with complete or partial response determined by a blinded independent review committee

SECONDARY OUTCOMES:
Objective response rate - Investigator assessment | Up to 24-months
  Percentage of patients with complete or partial response determined by the investigator
Complete response rate | Up to 24-months
  Percentage of patients who achieve a Complete Response determined by independent review committee and investigators assessment
Duration of response | Up to 24-months
  Duration of response (the time from the date of the first occurrence of complete response or partial response to the date of progression, relapse, or death from any cause) determined by independent review committee and investigators
Duration of complete response | Up to 24-months
  Time from the date of the first occurrence of CR to the date of progression, relapse, or death from any cause determined by independent review committee and investigators.
Progression-free survival | Up to 24-months
  Progression-free survival (the time from CRG-022 infusion until the first occurrence of disease progression or relapse) determined by independent review committee and investigator assessment
Overall Survival | Up to 24-months
  Overall Survival (the period from the date of CRG-022 infusion until the date of death from any cause) documented by the Investigator.
Incidence rate of adverse events | From Screening up to 15 years at protocol-defined timepoints
  Percentage of patients with treatment-related adverse events is assessed by CTCAEv5.0, CRS, ICANS, and IEC-HS graded by ASTCT criteria.

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - University of Arkansas Medical Sciences, Little Rock, Arkansas
  - City of Hope National Medical Center, Duarte, California
  - UCLA Division of Hematology Oncology, Los Angeles, California
  - Stanford University Hospital and Clinics, Stanford, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - University of Miami Hospital Sylvester Comprehensive Cancer Center, Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Northside Hospital, Atlanta, Georgia
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Iowa Hopitals & Clinics, Iowa City, Iowa
  - University of Kansas Medical Center Research Institute, Inc, Westwood, Kansas
  - University of Maryland Medical Center, Baltimore, Maryland
  - National Cancer Institute, Bethesda, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - New York University Medical Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Swedish Medical Center, Seattle, Washington
  - UW-Fred Hutchinson Cancer Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No